CLINICAL TRIAL: NCT03457220
Title: An Observational Study to Evaluate AZD9291 Treatment in Patients With EGFR T790M Positive Locally Advanced or Metastatic Non-small Cell Lung Cancer Following Progression on at Least One Prior EGFR TKI Treatment
Brief Title: An Observational Study to Evaluate AZD9291 Treatment in Patients With T790M Positive Non-small Cell Lung Cancer
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D5160R00021
Record Dates: First submitted 2018-03-01; First posted 2018-03-07 (Actual); Last update posted 2020-12-21 (Actual); Status verified 2020-12

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective

SUMMARY:
AZD9291 Early Access Program (EAP) was available in Taiwan during October 2015 to September 2016, a time period before the approval of AZD9291, to supply the unlicensed AZD9291 for the NSCLC patients who received at least one prior EGFR TKI therapy. At the end of September 2016, more than 450 patients have been under AZD9291 treatment through the EAP. This observational study aims to evaluate the clinical benefit of AZD9291 treatment for these patients who were in the EAP

DETAILED DESCRIPTION:
AZD9291 Early Access Program (EAP) was available in Taiwan during October 2015 to September 2016, a time period before the approval of AZD9291, to supply the unlicensed AZD9291 for the NSCLC patients who received at least one prior EGFR TKI therapy. At the end of September 2016, more than 450 patients have been under AZD9291 treatment through the EAP. This observational study aims to evaluate the clinical benefit of AZD9291 treatment for these patients who were in the EAP

ELIGIBILITY:
Inclusion Criteria:

* At least 20 years of age
* Patients who were in the AZD9291 Early Access Program
* Received at least one dose of AZD9291 treatment as mono-therapy, supported by available source documents
* Patient who discontinued the single use of AZD9291, had disease progression, or died under AZD9291 treatment, whichever comes last, during the period from October 01, 2015 to December 31, 2018
* Patients agree to provide the written informed consent or the informed consent is waived by IRB.

Exclusion Criteria:

• Patients who did not receive at least one dose of EGFR TKI for the treatment of EGFR mutation (+) NSCLC

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All the available patients who have participated in the AZD9291 EAP will be screened for the eligible criteria for data collection in this observational study
Sampling Method: Probability Sample
Enrollment: 423 (Actual)
Dates: Start 2018-06-21 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Progression free survival (PFS) | Every 12 weeks until treatment discontinuation as defined by RECIST 1.1 projected 12 months
  PFS is defined as the time interval (in months) from the first dose of AZD9291 in the EAP to the date of disease progression

SECONDARY OUTCOMES:
Overall survival (OS) | Every 12 weeks until treatment discontinuation as defined by RECIST 1.1 projected 24 months
  OS is defined as the time interval (in months) from the date of the first dose of AZD9291 in the EAP until the date of death due to any cause

OTHER OUTCOMES:
Response Rate (RR) | Every 12 weeks until treatment discontinuation as defined by RECIST 1.1 projected 12 months
  RR is defined as the percentage of subjects with the best overall response of 'responding', which is defined as complete response (CR) or partial response (PR), by investigator's assessment
Disease Control Rate (DCR) | Every 12 weeks until treatment discontinuation as defined by RECIST 1.1 projected 12 months
  DCR is defined as the percentages of subjects who have the best overall response of CR, PR, or SD, which is determined by investigator's assessment.
Time to treatment discontinuation (TTD) | Time from patient first dose to data cut off (up to 32 months)
  TTD is defined as the time interval (in months) from the date of the first dose of AZD9291 in the EAP until the date of the single use of AZD9291 discontinuation for any reason

CONTACTS AND LOCATIONS:
Locations (4):
- Taiwan (4):
  - Research Site, Kaohsiung City
  - Research Site, Taichung
  - Research Site, Tainan
  - Research Site, Taipei

REFERENCES:
- See also: CSR_Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5160R00021&attachmentIdentifier=d9ab5d4f-73bd-434e-9cb4-4205c318fd9e&fileName=D5160R00021_redacted_csr_synopsis.pdf&versionIdentifier=